CLINICAL TRIAL: NCT05740085
Title: Knowledge and Awareness of Osteoporosis in Rheumatoid Arthritis Patients
Brief Title: Osteoporosis Awareness in Rheumatoid Arthritis Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Uskudar State Hospital (Other Government)
Responsible Party: Principal Investigator, Mustafa Hüseyin Temel, Principal Investigator, Uskudar State Hospital
Other Study IDs: OPRA1
Record Dates: First submitted 2022-12-27; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Osteoporosis; Rheumatoid Arthritis
MeSH Terms: conditions — Osteoporosis; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rheumatoid Arthritis Patients: Patients that are diagnosed with rheumatoid arthritis
  Interventions: Other: Patient information form

INTERVENTIONS:
Other: Patient information form — Patients will be asked to fill out a patient information form and an osteoporosis awareness form

SUMMARY:
Osteoporosis is a condition that describes compromised skeletal microarchitecture in general, with clinical signs of decreased bone mineral density. Rheumatoid arthritis patients are at increased risk for developing osteoporosis. It is crucial to identify whether rheumatoid arthritis patients know and know about this disease. This study investigates awareness and knowledge of osteoporosis in rheumatoid arthritis patients.

DETAILED DESCRIPTION:
Osteoporosis is a common disease of bone loss. The reduced bone strength predisposes an increased risk for fractures in older individuals. It can affect people from different ethnicity. Many factors increase the risk of osteoporosis, including age, postmenopausal state, glucocorticoid use, low body weight, calcium, vitamin D, immobility, and chronic inflammation. Patients with rheumatoid arthritis are at high risk of developing osteoporosis due to chronic inflammation and the medications they use. Patients' knowledge and awareness about osteoporosis are essential for early detection, implementation of lifestyle changes, and treatment compliance. This study aimed to investigate osteoporosis awareness and knowledge about osteoporosis in patients with rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of rheumatoid arthritis
* Must be between the ages of 18 and 90
* Must give consent to participate in the study

Exclusion Criteria:

• Not giving consent

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 to 90 years with a diagnosis of rheumatoid arthritis who gave consent to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-04-30 (Estimated); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Level of knowledge in osteoporosis | 1 day
  Level of knowledge in osteoporosis will be assessed with revised osteoporosis knowledge test (OKT). The Revised OKT (2012) is a comprehensive instrument reflecting current research and assesses osteoporosis knowledge of adults. Responses offered to participants are multiple choice (e.g., for risk items: more likely, less likely, neutral, don't know), there is only one correct answer for each item. Responses are dichotomously recoded as correct or incorrect. In a U.S. sample of adults, the measure demonstrated internal consistency, very good stability, and content validity. Point-biserial correlations supported the measure's validity.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa H Temel, M.D., Study Chair — Uskudar State Hospital
Locations (1):
- Üsküdar State Hospital, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No